CLINICAL TRIAL: NCT00004253
Title: A Phase II Study of 3-Dimensional Conformal Hyperfractionation Radiation Therapy (3D-CHRT) With Dose Escalation and Amifostine Mucosal Protection for Patients With Favorable Prognosis Inoperable Stage II-IIIA/B Non-Small Cell Lung Cancer (NSCLC) Receiving Paclitaxel and Carboplatin
Brief Title: Combination Chemotherapy and Radiation Therapy in Treating Patients With Stage II or Stage III Non-small Cell Lung Cancer That Cannot Be Removed By Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Baptist Health South Florida (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067500; BHM-L1; BHM-99-64; NCI-V99-1582
Record Dates: First submitted 2000-01-28; First posted 2003-07-23 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2002-11

CONDITIONS: Lung Cancer
Keywords: stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Paclitaxel; Radiotherapy

INTERVENTIONS:
Drug: carboplatin
Drug: paclitaxel
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Specialized radiation therapy delivers a high dose of radiation directly to the tumor which may kill more tumor cells and cause less damage to normal tissue.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy and specialized high-dose radiation therapy in treating patients who have stage II or stage III non-small cell lung cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the probability of overall survival and local control in patients with favorable prognosis, unresectable stage II-IIIA/B non-small cell lung cancer receiving paclitaxel and carboplatin plus 3-D conformal hyperfractionation radiotherapy (3D-CHRT).
* Determine the incidence and severity of nonhematologic toxicity, specifically esophagitis and pneumonitis, during 3D-CHRT and chemotherapy with paclitaxel and carboplatin in these patients.
* Correlate complication rate with radiation based on the effective dose to determine safe treatment guidelines.
* Determine the feasibility of patient-specific dose escalation using this regimen in these patients.
* Determine the quality of life and symptom distress in these patients on this regimen.

OUTLINE: This is a dose-escalation study of 3-D conformal hyperfractionated radiotherapy (3D-CHRT).

Patients receive paclitaxel IV over 1 hour followed immediately by carboplatin IV over 30 minutes weekly for 6-8 weeks. Patients undergo 3D-CHRT twice daily five days a week for 6-8 weeks.

Cohorts of patients receive escalating doses of 3D-CHRT in 4 dose levels.

Quality of life is assessed prior to study, weekly during chemotherapy and radiotherapy, and at 3 and 6 months.

Patients are followed at 6 weeks, every 3 months for 1 year, every 6 months for 2 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 26-72 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patients with unresected locally advanced non-small cell lung cancer

  * Stage II, IIIA, or IIIB
  * No evidence of hematogenous metastases
* No pleural effusion(s) on chest x-ray (except after a thoracotomy or other invasive thoracic procedure)
* No intrathoracic tumor recurrence following resection

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 70-100%

Life expectancy:

* Not specified

Hematopoietic:

* Absolute granulocyte count at least 2,000/mm3
* Platelet count at least 130,000/mm3
* Hemoglobin at least 10 g/dL

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* SGOT no greater than 1.5 times upper limit of normal (unless caused by documented benign disease)

Renal:

* Creatinine no greater than 1.5 mg/dL

Cardiovascular:

* No active or symptomatic cardiac disease
* No acute myocardial infarction within the past 6 months
* No angina
* No congestive heart failure
* No uncontrolled arrhythmias
* Cardiac ejection fraction greater than 50%

Pulmonary:

* FEV1 at least 1.25 L AND
* DLCO at least 50% predicted

Other:

* Not pregnant
* Fertile patients must use effective contraception
* Weight loss no greater than 5% within 3 months of diagnosis
* No other prior malignancy within the past 3 years except nonmelanomatous skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior thoracic or neck radiotherapy

Surgery:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-03

CONTACTS AND LOCATIONS:
Overall Officials: Andre A. Abitbol, MD, Study Chair — Baptist Health South Florida
Locations (2):
- United States (2):
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida